CLINICAL TRIAL: NCT05939037
Title: Multicenter, Open-label, Phase II Study in Patients With Immunoglobulin M Monoclonal Gammopathy of Unknown Significance and Myelin Associated Glycoprotein Antibodies Related Polyneuropathy and Zanubrutinib Treatment - MAGNAZ Trial
Brief Title: Zanubrutinib Treatment in Patients With IgM Monoclonal Gammopathy and Antri-MAG Related Polyneuropathy
Acronym: MAGNAZ
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: BeiGene (Industry)
Responsible Party: Principal Investigator, Klaartje Nijssen, Principle Investigator, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22U-0179
Record Dates: First submitted 2023-05-23; First posted 2023-07-11 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Monoclonal Gammopathy of Uncertain Significance
MeSH Terms: conditions — Monoclonal Gammopathy of Undetermined Significance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Zanubrutinib Oral Product — Treatment will consist of Rituximab administered at 375 mg/m2 intravenously on Cycle 1 Days 1, 8, 15, 22 only (4 total infusions). The experimental part of the treatment will consist of Zanubrutinib, given once daily 320 mg (4 x 80 mg capsules). Although Zanubrutinib is taken continuously, therapy cycles are calculated per 28 days. Participants will be treated for a minimum of 6 cycles per protocol. Participants who still use Zanubrutinib at the end of study can continue indefinitely until registration and reimbursement in the Netherlands.

SUMMARY:
The objective of this investigator-initiated phase II single-arm open-label clinical trial is to investigate neurological response rate, safety and tolerability of Zanubrutinib 320 mg daily in combination with Rituximab 375 mg/m2 (standard therapy) for the treatment of immunoglobulin M monoclonal gammopathy of unknown significance (IgM MGUS) related polyneuropathy with Myelin Associated Glycoprotein antibodies (anti-MAG). 42 adult patients will be included in two Dutch hospitals (University Medical Center Utrecht and Amsterdam University Medical Center). This trial consists of a 6-month treatment period, after which the hematological response will be evaluated. Adequately responding participants (at least partial response) will be treated for an additional 6 months, after which hematological response will be re-evaluated. Participants with at least a very good partial response will remain on treatment. Non-responding participants will be followed for clinical outcomes only. The total study period per participant will be 36 months.

DETAILED DESCRIPTION:
SYNOPSIS Multicenter, open-label, phase II study in patients with immunoglobulin M monoclonal gammopathy of unknown significance and Myelin Associated Glycoprotein antibodies related polyneuropathy and Zanubrutinib Treatment - MAGNAZ trial

Rationale Polyneuropathy (PNP) associated with immunoglobulin M (IgM) monoclonal gammopathy of unknown significance (MGUS) and myelin associated glycoprotein (MAG) antibodies (IgM MGUS/anti-MAG PNP) is characterized by severe sensory dysfunction, ataxia, imbalance, tremor and distal weakness of the arms and legs. It is a chronic and progressive PNP that leads to significant disability. The IgM M-protein that is produced by the MGUS B-cell clone has anti-MAG properties, and treatment options are aimed at lowering the M protein level. Treatment response is associated with a decrease in M-protein and anti-MAG antibodies. At present, the only treatment option is Rituximab (an anti-cluster of differentiation antigen 20 (CD20) monoclonal antibody), which effectuates a limited but clinically meaningful neurological improvement in approximately 30% of patients.

IgM MGUS/anti-MAG PNP shares in many cases the same genetic mutation in the MYD88 gene as seen in Waldenström's Macroglobulinemia (WM). This mutation is associated with an enhanced sensitivity to a novel type of drugs: Bruton's Tyrosine Kinase (BTK) inhibitors. WM patients have recently been successfully treated with BTK inhibitors. One of these BTK inhibitors, Zanubrutinib, has been given to many patients with hematological malignancies and is considered a safe drug. In WM, Zanubrutinib lowers the IgM levels with minimal 50% in 77% of patients. It has been approved for several malignancies in Europe and the USA. Importantly, and in contrast to other drugs, chemotherapy induced PNP is not a side effect. Considering the genetic link between IgM MGUS/anti-MAG PNP and WM, the investigators postulate that BTK-inhibitors are also able to effectively treat IgM MGUS/anti-MAG PNP and alleviate the severe neurological symptoms.

Objective The investigators want to investigate the use of Zanubrutinib in combination with standard therapy Rituximab for the possible improvement on the neurological outcome in patients with IgM MGUS/anti-MAG PNP. In addition, the investigators want to investigate safety and tolerability of this treatment.

Main trial endpoints As main endpoints, the investigators aim to explore initial improvement of neurological disability after 12 months and safety and tolerability of Zanubrutinib treatment. For the neurological primary endpoint, neurological disability will be measured with the Inflammatory Neuropathy Cause and Treatment (INCAT) disability score. The investigators will use proportion of patients with ≥2 points improvement on the INCAT disability score as primary endpoint. For safety and tolerability, the investigators will determine the rate of treatment related adverse events classified according to the Medical Dictionary for Regulatory Activities and graded according to the Common Terminology Criteria for Adverse Events version 5.0 and dose changes, and the investigators will evaluate adherence to Zanubrutinib by counting early withdrawals.

Secondary trial endpoints Secondary endpoints include patient reported outcome measures (PROM's) and other neurological function measurements and hematological response rate. In addition, the investigators will evaluate molecular mutations and the change in anti MAG titers.

Trial design This is an investigator-initiated, phase 2a, single-arm, open-label clinical trial to investigate whether the combined treatment of Zanubrutinib and Rituximab can be a potentially beneficial treatment of IgM MGUS/anti-MAG PNP, what the expected effect size of this treatment on IgM MGUS/anti-MAG PNP is to possibly inform a larger randomized controlled trial, and whether this treatment is safe and tolerable. In total, 2 hospitals in the Netherlands will participate to enroll 42 patients. The accrual period will consist of 1 year. The study will consist of a 6-month treatment period, after which the hematological response will be evaluated. Adequately responding participants (at least partial response) will be treated for an additional 6 months, after which hematological response will be re-evaluated. Participants with at least a very good partial response will remain on treatment. Non-responding participants will be followed for clinical outcomes only. The total study period per participant will be 36 months. participants will visit the clinic every month during the first 6 months, every 2 months during the subsequent 6 months and every 3 months during the follow-up period. Each visit will take approximately 1 hour.

Trial population Patients of 18 years and older with established IgM MGUS/anti-MAG PNP following the standard criteria may be eligible for the trial. All patients must have signed an informed consent to be registered before start of treatment and must meet all eligibility criteria.

Interventions Treatment Treatment will consist of Rituximab administered at 375 mg/m2 intravenously on Cycle 1 Days 1, 8, 15, 22 only (4 total infusions). The experimental part of the treatment will consist of Zanubrutinib, given once daily 320 mg (4 x 80 mg capsules). Although Zanubrutinib is taken continuously, therapy cycles are calculated per 28 days. Participants will be treated for a minimum of 6 cycles per protocol. Participants who still use Zanubrutinib at the end of study can continue indefinitely until registration and reimbursement in the Netherlands.

Diagnostic procedures At the first visit, the investigators will screen for trial eligibility, which includes a bone marrow aspiration and biopsy, electrocardiogram (ECG), medical history inquiry including prior medicine usage, physical examination, neurological examination including questionnaires, urine analysis, pregnancy test and blood tests. Every visit, the investigators will obtain a blood sample to measure the pharmacodynamic response and monitor treatment safety. Additionally, the investigators will perform physical examinations and neurological examinations (including questionnaires) to monitor treatment effect.

Ethical considerations relating to the clinical trial including the expected benefit to the individual participant or group of patients represented by the trial participants as well as the nature and extent of burden and risks This trial investigates the potential positive effect of Zanubrutinib on a severe progressive neurological disease by lowering the disease-causing IgM M protein. For this disabling disease there is currently limited effective treatment. Zanubrutinib is an approved medicine that has been used for associated hematological malignancies such as WM. Side effects are regarded acceptable. Potential benefits are on the individual level, which is reflected by one of the main endpoints that reflects neurological functional improvement. Since this trial investigates Zanubrutinib treatment for a disease wherein it is not approved at present, the investigators will closely monitor safety and response by means of frequent blood analyses and outpatient clinic visits.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent and understand and comply with the requirements of the study
* Demyelinating PNP defined by the European Federation of Neurological Societies/Peripheral Nerve Society guideline on management of paraproteinemic demyelinating neuropathies (84)
* Functional impairment; defined as an INCAT disability score (INCATds) of ≥2
* Age ≥ 18 years
* IgM MGUS, defined as the presence of an IgM M-protein (detectable but < 30 g/L) AND elevated total IgM level in serum
* Presence of anti MAG antibodies ≥ 10.000 titer units, measured with the Bühlmann ELISA
* Eastern Cooperative Oncology Group (ECOG) performance score 0, 1, or 2 (85)
* Adequate hematological laboratory values defined as hemoglobin ≥ 6.0 mmol/L, neutrophils > 1.0 × 109/L and platelets > 100 × 109/L
* Adequate hepatic and renal function laboratory values defined as aspartate transaminase (ASAT)/ alanine aminotransferase (ALAT) < 3 × upper limit of normal (ULN), bilirubin < 1.5× ULN and creatinine clearance ≥ 30 ml/min
* Patients with hypertension can only be enrolled when blood pressure is adequately treated, defined as systolic blood pressure of <140 mmHg and diastolic blood pressure of <90 mmHg at screening
* No history of severe bleeding disorder such as hemophilia A, hemophilia B, von Willebrand disease, or history of spontaneous bleeding requiring blood transfusion or other medical intervention
* Previous treatment with intravenous immunoglobulins is allowed if > 3 months before inclusion
* Previous treatment for PNP with Anti CD20 monoclonal antibody (MoAb) and/or cyclophosphamide is allowed only if given > 6 months before inclusion. Patients without previous response to Rituximab >6 months before inclusion can be included.

Exclusion Criteria:

* Hematological malignancy e.g., known Multiple Myeloma or confirmed Waldenström's Macroglobulinemia based on bone marrow analysis
* Any history of malignancy of any organ system (other than localized basal or squamous cell carcinoma of the skin, superficial bladder cancer or carcinoma in situ of the cervix or breast), treated or untreated within the last 3 years
* History of ischemic stroke within 180 days before first dose of Zanubrutinib
* History of central nervous system (CNS) hemorrhage
* History of inherited or acquired hemorrhagic disorder
* Prior treatment with purine analogues (fludarabine or cladribine)
* Prior treatment with a BTK inhibitor
* Major surgery within 4 weeks of study treatment
* Participation in another interventional clinical trial
* Pregnant women, women with child-bearing potential (WOCBP) not able or willing to prevent pregnancy and lactating women as well. WOCBP will agree to use highly effective contraception for the duration of the trial treatment and for 12 months after Rituximab treatment stop or 120 days after Zanubrutinib treatment stop, whichever has a longer duration. Participants using hormonal contraceptives (e.g., birth control pills or devices) must use a barrier method of contraception (e.g., condoms) as well.
* Other known concomitant causes of chronic (demyelinating) PNP, including Charcot Marie Tooth Disease, other hereditary neuropathies, diabetes mellitus, use of amiodarone, past or current dependence on alcohol, other lymphoma or malignant blood dyscrasias, previous Guillain-Barré syndrome
* Currently active, clinically significant cardiovascular disease such as uncontrolled arrhythmia, congestive heart failure, any Class 3 or 4 cardiac disease (congestive heart failure) as defined by the New York Heart Association (NYHA) Functional Classification, or history of myocardial infarction within 6 months of screening
* A history of clinically significant ECG abnormalities, or any of the following ECG abnormalities at screening:

  * The corrected QT interval by Fridericia (QTcF) >450 msec (males)
  * QTcF >460 msec (females)
  * History of familial long QT syndrome or known family history of Torsade de Pointes
  * Use of agents known to prolong the QT interval unless they can be permanently discontinued for the duration of the study
  * Second degree atrioventricular (AV) block Type II, or third-degree AV block
  * Controlled atrial fibrillation is allowed
* Unable to swallow capsules or disease significantly affecting gastrointestinal function such as malabsorption syndrome, resection of the stomach or small bowel, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction
* Uncontrolled active systemic infection or recent infection requiring parenteral anti-microbial therapy that was completed ≤ 14 days before the first dose of study drug. Active tuberculosis.
* Infection with human immunodeficiency virus (HIV), or serologic status reflecting active hepatitis B or hepatitis C infection. Patients with presence of hepatitis C virus (HCV) antibody are eligible if HCV ribonucleic acid (RNA) is undetectable. Patients with a serologic status reflecting prior or active hepatitis B cannot be included. We will test the hepatitis B surface antigen (HBsAg), anti-hepatitis B core antibodies (anti-HBc) and anti-hepatitis B surface antibodies (anti-HBs) at screening. Patients with a serological status reflecting an earlier hepatitis B vaccination (HBsAg negative / antiHBc negative / anti-HBs positive) may be included. Other combinations are not allowed.
* At time of study entry, taking any medications which are strong Cytochrome P450, family 3, subfamily A (CYP3A) inhibitors (e.g., conivaptan, posaconazole, voriconazole, ketoconazole, itraconazole, clarithromycin, indinavir, lopinavir, ritonavir, telaprevir) or strong CYP3A inducers (e.g., carbamazepine, phenytoin, rifampin, St. John's wort)
* Intolerance to previous Rituximab treatment
* History of intolerance to the active ingredients or other ingredients of Zanubrutinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with ≥2 points improvement on the INCAT disability score | At the end of Cycle 12 (each cycle is 28 days)
  To assess the improvement of the functional neurological outcome of participants after treatment with Zanubrutinib in combination with Rituximab by The Inflammatory Neuropathy Cause and Treatment (INCAT) disability score (Overall score is the sum of arm and leg disability, scaled 0 (no problems) to 5 (disabled).
  A proportion of patients with ≥2 points improvement on the INCAT disability score wil be used as primary endpoint
Incidence of adverse events during treatment and follow up by the Common Terminology Criteria for Adverse Events (CTCAE), version 5 | Till 36 months from baseline
  To assess the safety and tolerability of the combined treatment with Rituximab and Zanubrutinib
Study Drug adherence | Till end of treatment, which will be after 6 or 12 cycles (each cycle is 28 days)
  Dose adjustments made per patient.Registration of drug accountability (counting of remaining capsules after each treatment cycle). Drug accountability will be presented as percentage.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Utrecht, Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided